CLINICAL TRIAL: NCT02627274
Title: An Open-Label, Multicenter, Dose-Escalation, Phase Ia/Ib Study to Evaluate Safety, Pharmacokinetics, and Therapeutic Activity of RO6874281, an Immunocytokine Consisting of Interleukin 2 Variant (IL-2v) Targeting Fibroblast Activation Protein-α (FAP), as a Single Agent (Part A) or in Combination With Trastuzumab or Cetuximab (Part B or C)
Brief Title: A Study Evaluating Safety, Pharmacokinetics, and Therapeutic Activity of RO6874281 as a Single Agent (Part A) or in Combination With Trastuzumab or Cetuximab (Part B or C)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP29842; 2015-002251-97 (EudraCT Number)
Record Dates: First submitted 2015-11-26; First posted 2015-12-10 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumor; Breast Cancer; Cancer of Head and Neck
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms | interventions — Trastuzumab; Cetuximab

ARMS (3):
- Part A: RO6874281 Monotherapy (Experimental): Dose Escalation: RO6874281 will be administered as an intravenous (IV) infusion. The starting dose regimen of RO6874281 as a single agent will be 5 milligrams (mg) once weekly (QW). Different regimens may be explored based on the emerging safety, PK, and PD data of RO6874281 and may be tested in parallel. Participants will be treated with RO6874281 until disease progression, unacceptable toxicities, or withdrawal of consent. Participants may continue treatment with RO6874281 for a maximum of 24 months.
  Interventions: Drug: RO6874281
- Part B: RO6874281 in Combination with Trastuzumab (Experimental): Dose Escalation: RO6874281 will be administered as an IV infusion. RO6874281 will be administered QW for the first 4 administrations, then Q2W. The standard dose for trastuzumab will be a loading dose of 6 milligrams per kilogram (mg/kg) followed by a maintenance dose of 4 mg/kg from Cycle 2 in a Q2W regimen. Different regimens may be explored based on the emerging safety, PK, and PD data of RO6874281 and may be tested in parallel. Participants will be treated with RO6874281 in combination with trastuzumab until disease progression, unacceptable toxicities, or withdrawal of consent. Participants may continue treatment with RO6874281 in combination with trastuzumab for a maximum of 24 months.
  Interventions: Drug: RO6874281; Drug: Trastuzumab
- Part C: RO6874281 in Combination with Cetuximab (Experimental): RO6874281 will be administered as an IV infusion. The starting dose regimen of RO6874281 in combination with cetuximab will be 5 mg QW for the first 4 administrations, then Q2W. Cetuximab will be administered Q2W at 500 milligrams per square meter (mg/m^2). Different regimens may be explored based on the emerging safety, PK, and PD data of RO6874281 and may be tested in parallel. Participants will be treated with RO6874281 in combination with cetuximab until disease progression, unacceptable toxicities, or withdrawal of consent. Participants may continue treatment with RO6874281 in combination with cetuximab for a maximum of 24 months.
  Extension Phase: The MTD for RO6874281 was determined to be 10mg and therefore patients in the extension will be treated with 10mg RO6874281. Cetuximab and R06874281 will be administered weekly during induction phase (cycle 1 and cycle 2). Both IMPs will be administered Q2W starting in cycle 3.
  Interventions: Drug: RO6874281; Drug: Cetuximab

INTERVENTIONS:
Drug: RO6874281 — RO6874281 will be administered as per the schedule specified under arm description.
  Other Names: simlukafusp alfa
Drug: Trastuzumab — Trastuzumab will be administered as per the schedule specified under arm description.
  Other Names: Herceptin
  Arms: Part B: RO6874281 in Combination with Trastuzumab
Drug: Cetuximab — Cetuximab will be administered as per the schedule specified under arm description.
  Arms: Part C: RO6874281 in Combination with Cetuximab

SUMMARY:
This first-in-human, open-label, multicenter, Phase Ia/Ib, adaptive, multiple ascending-dose study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary anti-tumor activity of RO6874281 as a single agent (Part A) or in combination with trastuzumab or cetuximab (Part B or C).

ELIGIBILITY:
Inclusion Criteria:

* Radiologically measurable and clinically evaluable disease
* Absence of rapid disease progression or threat to vital organs or critical anatomical sites requiring urgent alternative medical intervention
* Confirmed at least one tumor lesion with location accessible to safely biopsy per clinical judgment (special requirements apply for Part C; Participants with only one target lesion and no non-target lesions can enroll after documented agreement with the Medical Monitor).
* Life expectancy of greater than or equal to (>=12) weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Participants with unilateral pleural effusion (other than non-small cell lung cancer [NSCLC] indication) should fulfill the following criteria for pulmonary and cardiac functions: Global Initiative for Chronic Obstructive Lung Disease (GOLD) classification 0 - 1 level and New York Heart Association (NYHA) classification class 1 or better
* Forced expiratory volume 1 (FEV1) >70% and forced vital capacity (FVC) >70% of predicted value; participants with lung metastases should present with DLCO >60% of predicted value
* Adequate cardiovascular, hematological, liver and renal function
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to grade less than or equal to (<=) 1, except alopecia (any grade) and Grade 2 peripheral neuropathy
* Negative serum pregnancy test within 7 days prior to study treatment in premenopausal women and women less than (<) 12 months after menopause
* For women who are not postmenopausal and have not undergone surgical sterilization: agreement to remain abstinent or use two adequate non-hormonal methods of contraception, including at least one method with a failure rate of <1 percent (%) per year, during the treatment period and for a period of time after the last dose of study drug(s) as defined in the protocol
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm during the treatment period and for at least for at least 2 months after the last dose of study treatment
* For Part A exclusively (RO6874281 monotherapy), confirmed advanced and/or metastatic solid tumor, with at least one tumor lesion of location accessible to biopsy per clinical judgment of the treating physician, and confirmed progression at baseline; for whom no standard therapy that would confer clinical benefit to the participant exists
* For Part B exclusively (RO6874281 in combination with trastuzumab), participants with metastatic or recurrent or locally advanced human epidermal growth factor receptor 2 (HER2)-positive breast cancer, as defined by the College of American Pathologists HER2 testing guidelines, who have progressed on at least two lines of HER2-directed therapies in the metastatic setting and the last therapy prior to going on study has to contain a HER2-directed antibody; baseline left ventricular ejection fraction (LVEF) of >=50% (measured by echocardiography) predose on Cycle 1 Day 1
* For Part C exclusively (RO6874281 in combination with cetuximab), participants with recurrent, unresectable or metastatic squamous cell carcinoma of the head and neck. Participants can have had standard or experimental treatment, including but not limited to radiation therapy, chemotherapy, or immunotherapy
* Participants with Gilbert's syndrome will be eligible for the study

Exclusion Criteria:

* History of, active, or suspicion of autoimmune disease (exceptions apply)
* Adverse events from prior anti-cancer therapy that have not resolved to Grade 1, except for alopecia, vitiligo, or endocrinopathies managed with replacement therapy
* Symptomatic or untreated central nervous system (CNS) metastases
* History of treated asymptomatic CNS metastases with any of the following: Metastases to the brain stem, midbrain, pons, medulla, cerebellum, or within 10 millimeters (mm) of the optic nerves and chiasm; history of intracranial or spinal cord hemorrhage; lacking radiographic demonstration of improvement upon the completion of CNS-directed therapy and evidence of progression between completion of therapy and the baseline radiographic study; ongoing requirement for dexamethasone; stereotactic or whole brain radiation within 28 days before the start of study treatment; last CNS radiographic study less than 4 weeks since completion of radiotherapy and less than 2 weeks since the discontinuation of corticosteroids; CNS metastases treated by resection or brain biopsy performed within 28 days before the start of study treatment
* Participants with an active second malignancy
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders, and known autoimmune diseases or other disease with ongoing fibrosis
* Participants (all indications) with confirmed bilateral pleural effusion and NSCLC participants with confirmed uni- or bilateral pleural effusion by X-ray are not eligible
* Significant cardiovascular/cerebrovascular disease within 6 months prior to Day 1 of study drug administration
* Active or uncontrolled infections
* Known human immunodeficiency virus (HIV) or known active hepatitis B virus or hepatitis C virus infection
* History of chronic liver disease or evidence of hepatic cirrhosis
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that give reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury <28 days prior to the first RO6874281 infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Dementia or altered mental status that would prohibit informed consent
* Pregnant or breastfeeding women
* Known hypersensitivity to any of the components of RO6874281
* Concurrent therapy with any other investigational drug
* Immune-related endocrinopathies
* Immunomodulating agents <28 days prior to first dose of study drug
* Treatment with systemic immunosuppressive medications
* Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy
* For Part B exclusively, known hypersensitivity to any of the components of trastuzumab
* For Part C exclusively, known hypersensitivity to any of the components of cetuximab
* For Parts A, B, and C, eligibility of participants who require blood transfusion before and after the start of the study treatment should be discussed by the Sponsor and investigator
* For Parts B and C, Participant eligibility for treatment with trastuzumab or cetuximab should be verified against trastuzumab or cetuximab labeling documents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 21
Maximum Tolerated Dose (MTD) of RO6874281 | Day 1 up to Day 21
Optimal Biological Dose (OBD) of RO6874281 | Day 1 up to Day 21
Recommended Dose for Further Development of RO6874281 | Day 1 up to Day 21
Systemic Clearance (CL) of RO6874281 | Day 1 up to 24 months
Volume of Distribution at Steady State (Vss) of RO6874281 | Day 1 up to 24 months
Area Under the Concentration-Time Curve (AUC) of RO6874281 | Day 1 up to 24 months
Maximum Observed Serum Concentration (Cmax) of RO6874281 | Day 1 up to 24 months

SECONDARY OUTCOMES:
Number of T Cells in the Peripheral Blood | Day 1 up to 24 months
Number of Natural Killer (NK) Cells in the Peripheral Blood | Day 1 up to 24 months
Density of Cluster of Differentiation (CD)8+ Cells in Tumor Samples | Day 1 up to 24 months
Density of CD3-/Perforin+ Cells in Tumor Samples | Day 1 up to 24 months
Density of CD20 Cells in Tumor Samples | Day 1 up to 24 months
Percentage of Participants With Overall Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Day 1 up to 24 months
Percentage of Participants With Disease Control According to RECIST v1.1 | Day 1 up to 24 months
Progression-Free Survival (PFS) According to RECIST v1.1 | Day 1 up to 24 months
Percentage of Participants With Overall Response According to Modified RECIST | Day 1 up to 24 months
Percentage of Participants With Disease Control According to Modified RECIST | Day 1 up to 24 months
PFS According to Modified RECIST | Day 1 up to 24 months
Percentage of Participants With Overall Response According to iRECIST | Day 1 up to 24 months
Percentage of Participants With Disease Control According to iRECIST | Day 1 up to 24 months
PFS According to iRECIST | Day 1 up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (5):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UCSD - Moores Cancer Center, La Jolla, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Washington University; Division of Oncology, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
- UZ Antwerpen, Edegem, Belgium
- Canada (2):
  - Juravinski Cancer Clinic; Department of Oncology, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- France (5):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Sitep, Villejuif
- Italy (5):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Fondazione IRCCS Istituto Nazionale dei Tumori;S.S. Trattamento MedicoTumori dellaTesta e delCollo, Milan, Lombardy
  - Istituto Europeo di Oncologia; Svil. Nuovi Farmaci per Terapie Innovative, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda); Oncologico -Onc.Falck, Milan, Lombardy
  - Ospedale Policlinico S. Matteo; Phase I Clinical Trial Unit and Experimental Therapy, Pavia, Lombardy
- Netherlands (2):
  - Antoni Van Leeuwenhoek Ziekenhuis; Gastro-Enterologie, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (2):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Christie Hospital, Manchester

REFERENCES:
- [Derived] Hansen AR, Gomez-Roca CA, Robbrecht DGJ, Verlingue L, Italiano A, Bauman JE, Steeghs N, Prenen H, Fayette J, Spicer J, Niu J, Habigt C, Schneider M, Evers S, Sleiman N, Dejardin D, Ardeshir C, Schmid D, Boetsch C, Charo J, Kraxner A, Teichgraber V, Keshelava N, Bonomi MR. Phase Ib Study of the Immunocytokine Simlukafusp Alfa (FAP-IL2v) in Combination with Cetuximab in Patients with Head and Neck Squamous Cell Carcinoma. Clin Cancer Res. 2024 Dec 16;30(24):5540-5547. doi: 10.1158/1078-0432.CCR-24-1562. PMID 39422604